CLINICAL TRIAL: NCT00534599
Title: A Multicenter, Rand., Double-blind, Parallel-group, Pbo-controlled Study of the Efficacy and Safety of SEROQUEL® XR Compared With Pbo as an Adjunct to Treatment in Patients With Generalized Anxiety Disorder Who Demonstrate Partial or No Response to a SSRI or SNRI Alone or in Combination With a Benzo
Brief Title: Generalized Anxiety Disorder Adjunct Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1441L00016
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Results first posted 2011-04-05 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Anxiety; Anxiety Disorders; Anxiety Neuroses; Anxiety States
Keywords: Generalized anxiety disorders; anxiety; adjunct treatment in anxiety; anxiety disorder; partial or non-responder in anxiety
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Other): Adjunctive Placebo Seroquel XR to anxiety treatment
  Interventions: Drug: Placebo
- 2 (Experimental): Adjunctive Seroquel XR to anxiety treatment
  Interventions: Drug: quetiapine fumarate XR

INTERVENTIONS:
Drug: Placebo — oral
  Arms: 1
Drug: quetiapine fumarate XR — oral
  Other Names: Seroquel XR
  Arms: 2

SUMMARY:
This study is being carried out to see if extended release quetiapine fumarate (Seroquel®XL) when added to standard selective serotonin reuptake inhibitor (SSRI) / serotonin-norepinephrine reuptake inhibitor (SNRI) therapy is effective and safe for the treatment of Generalized Anxiety Disorder in patients with partial or no response to SSRI/SNRI alone or in combination with a benzodiazepine, and if so, how it compares with placebo

ELIGIBILITY:
Inclusion Criteria:

Provision of Informed Consent

* Documented diagnosis of Generalized Anxiety Disorder
* Female patients must not be pregnant and be willing to use a reliable method of birth control
* Be able to understand and comply with study requirements

Exclusion Criteria:

Other psychiatric disorders that could confound the study results, as judged by the study doctor

* Moderate to severe depression
* Other clinically relevant diseases, as judged by the study doctor
* Medication that you are taking, as judged by the study doctor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Brecher, MD, Study Director — AstraZeneca
Locations (53):
- United States (53):
  - Research Site, Birmingham, Alabama
  - Research Site, Little Rock, Arkansas
  - Research Site, Beverly Hills, California
  - Research Site, Encino, California
  - Research Site, Fresno, California
  - Research Site, La Mesa, California
  - Research Site, Oceanside, California
  - Research Site, Redlands, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Sherman Oaks, California
  - Research Site, Bradenton, Florida
  - Research Site, Dayton, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Maitland, Florida
  - Research Site, Miami, Florida
  - Research Site, North Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Lafayette, Indiana
  - Research Site, Merrillville, Indiana
  - Research Site, Terre Haute, Indiana
  - Research Site, Prairie Village, Kansas
  - Research Site, Owenboro, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Rockville, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Cherry Hill, New Jersey
  - Research Site, Clementon, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Cedarhurst, New York
  - Research Site, Fresh Meadows, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Staten Island, New York
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Salem, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Witchita Falls, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington

REFERENCES:
- [Derived] Khan A, Atkinson S, Mezhebovsky I, She F, Leathers T, Pathak S. Extended-release quetiapine fumarate (quetiapine XR) as adjunctive therapy in patients with generalized anxiety disorder and a history of inadequate treatment response: a randomized, double-blind study. Ann Clin Psychiatry. 2014 Feb;26(1):3-18. PMID 24660224
- [Derived] Khan A, Atkinson S, Mezhebovsky I, She F, Leathers T, Pathak S. Extended-release quetiapine fumarate (quetiapine XR) as adjunctive therapy in patients with generalized anxiety disorder and a history of inadequate treatment response: a randomized, double-blind study. Ann Clin Psychiatry. 2013 Nov;25(4):E7-22. PMID 24199224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient enrollment from 31 August 2007 to 02 September 2008
Pre-assignment Details: Wash-out period of up to 35 days for discontinuation of prohibited medications
Groups:
- Quetiapine XR: 50 mg to 300 mg extended release tablets once daily
- Placebo: Matching placebo tablets once daily
Period: Overall Study
Arm/Group | Quetiapine XR | Placebo
Started | 209 (Randomized) | 200 (Randomized)
Completed | 152 | 168
Not Completed | 57 | 32
Not completed — Adverse Event | 25 | 4
Not completed — Incorrect enrollment | 2 | 1
Not completed — Mis-randomization | 2 | 2
Not completed — Developed study-specific d/c criteria | 5 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Generalized anxiety disorder worsened | 0 | 1
Not completed — Protocol Violation | 1 | 3
Not completed — Lost to Follow-up | 11 | 14
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Other | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine XR | Placebo | Total
Number analyzed (Participants) | 204 | 198 | 402
Age Continuous [Mean (Standard Deviation); unit: Years] | 46.6 (12.1) | 44.2 (10.9) | 44.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 150 | 296
  Male | 58 | 48 | 106

OUTCOME MEASURES:

1. Primary Outcome: Least Square Mean Change From Randomization to Week 8 in Hamilton Rating Scale for Anxiety (HAM-A) Total Score
Description: Hamilton Rating Scale for Anxiety (HAM-A) consists of 14 items to evaluate anxiety. Each item is rated on a scale from 0-4, with '0' showing no anxiety (not present) and '4' showing the worst (very severe).
  Results based on MITT population with available data for this outcome measure. Least square mean of each treatment was adjusted for baseline value.
Time Frame: Baseline (randomization) and then 8 weeks
Population: Results participant numbers are based on Modified Intention to Treat (MITT) population set; The participants in the overall study are participants randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 204 | 198
units on scale | -10.74 [-12.01 to -9.47] | -9.61 [-10.89 to -8.32]

2. Secondary Outcome: Least Square Mean Change From Randomization to Week 8 in Clinical Global Impression-Severity of Illness (CGI-S) Score
Description: The CGI-S is assessed on a seven-point scale ranging from most extremely ill/very much worse (7) to normal/very much improved (1).
  Results based on MITT population with available data for this outcome measure.
Time Frame: Baseline (randomization) and then 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: LS mean change from randomization
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 204 | 198
LS mean change from randomization | -1.36 [-1.56 to -1.15] | -1.13 [-1.34 to -0.93]

3. Secondary Outcome: Number of Patients With Clinical Global Impression-Global Improvement (CGI-I) Score of "Much/Very Much Improved" at Week 8
Description: This pertains to the CGI-I scale which rates improvement of anxiety on a scale from 1-7, with '1' showing the best improvement(Very Much Improved) and '7' showing the worst improvement (Very Much Worse) as compared to the baseline visit. A rating of '2' indicates 'Much Improved'.
  Results based on MITT population with available data for this outcome measure.
Time Frame: Baseline (randomization) and then 8 weeks
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 204 | 198
Participants | 114 | 97

4. Secondary Outcome: Least Square Mean Change From Randomization to Week 8 in HAM-A Psychic Anxiety Subscale Score
Description: The HAM-A psychic anxiety factor subscale is defined as the sum of the following 7 HAM-A factors: anxious mood, tension, fears, insomnia, intellectual, depressed mood and behavior at the interview (i.e.items 1-6 and 14, respectively) Results based on MITT population with available data for this outcome measure.
Time Frame: Baseline (randomization) and then 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: LS mean change from randomization
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 204 | 198
LS mean change from randomization | -6.09 [-6.81 to -5.37] | -5.21 [-5.94 to -4.49]

5. Secondary Outcome: Least Square Mean Change From Randomization to Week 8 in HAM-A Somatic Anxiety Subscale Score
Description: The HAM-A Somatic cluster subscale is defined as the sum of the following 7 HAM-A items: somatic (muscular), somatic (sensory), cardiovascular symptoms, respiratory symptoms, gastrointestinal symptoms, genitourinary symptoms and autonomic system (i.e. items 7-13 respectively).
  Results based on MITT population with available data for this outcome measure.
Time Frame: Baseline (randomization) and then 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: LS mean change from randomization
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 204 | 198
LS mean change from randomization | -4.63 [-5.25 to -4.02] | -4.38 [-5.0 to -3.75]

6. Secondary Outcome: Number of Patients With HAM-A Response (≥50% Score Reduction From Randomization) at Week 8
Description: Hamilton Rating Scale for Anxiety (HAM-A) response is derived from the HAM-A total score and is defined as a decrease from baseline total HAM-A score of at least 50%. (1=Yes, 0=No) Results based on MITT population with available data for this outcome measure.
Time Frame: Baseline (randomization) and then 8 weeks
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 204 | 198
Participants | 84 | 72

7. Secondary Outcome: Number of Patients With HAM-A Remission (Total Score ≤7) at Week 8
Description: Hamilton Rating Scale for Anxiety (HAM-A) remission is derived from the HAM-A total score and is defined as a HAM-A total score of ≤7. 1=Yes, 0=No Results based on MITT population with available data for this outcome measure.
Time Frame: Baseline (randomization) and then 8 weeks
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 204 | 198
Participants | 48 | 34

8. Secondary Outcome: Least Square Mean Change From Randomization to Week 8 in Quality of Life Enjoyment and Satisfaction Questionaire (Q-LES-Q) Percent Maximum Total Score
Description: The Q-LES-Q score is the sum of the first 14 items, larger values indicating a higher perceived quality of life enjoyment and satisfaction. This total score was converted to a % maximum score using the following scoring conversion: %Maximum score = (Total score-14)*(100/560)rounded to an integer.
  Results based on MITT population with available data for this outcome measure.
Time Frame: Baseline (randomization) and then 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: LS mean change from randomization
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 202 | 194
LS mean change from randomization | 7.33 [5.4 to 9.26] | 6.43 [4.46 to 8.40]

9. Secondary Outcome: Mean Change From Randomization to Week 8 in Q-LES-Q Item 15 (Satisfaction With Medication) Score
Description: Results based on MITT population with available data for this outcome measure.
Time Frame: Baseline (randomization) and then 8 weeks
Measure: Mean (Standard Deviation); unit: Mean change from randomization
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 179 | 174
Mean change from randomization | 0.30 (1.10) | 0.40 (1.10)

10. Secondary Outcome: Mean Change From Randomization to Week 8 in Q-LES-Q Item 16 (Overall Quality of Life) Score
Description: Results based on MITT population with available data for this outcome measure.
Time Frame: Baseline (randomization) and then 8 weeks
Measure: Mean (Standard Deviation); unit: Mean change from randomization
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 204 | 198
Mean change from randomization | 0.30 (1.0) | 0.20 (0.90)

11. Secondary Outcome: Least Square Mean Change From Randomization to Week 1 in HAM-A Total Score
Description: Hamilton Rating Scale for Anxiety (HAM-A) consists of 14 items to evaluate anxiety. Each item is rated on a scale from 0-4, with '0' showing no anxiety (not present) and '4' showing the worst (very severe).
  Results based on MITT population with available data for this outcome measure.
Time Frame: Baseline (randomization) and then 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: LS mean change from randomization
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 195 | 191
LS mean change from randomization | -6.45 [-7.50 to -5.41] | -4.47 [-5.52 to -3.41]

12. Secondary Outcome: Least Square Mean Change From Randomization to Week 1 in HAM-A Psychic Anxiety Subscale Score
Description: Hamilton Rating Scale for Anxiety (HAM-A) consists of 14 items to evaluate anxiety. Each item is rated on a scale from 0-4, with '0' showing no anxiety (not present) and '4' showing the worst (very severe).Results based on MITT population with available data for this outcome measure.
Time Frame: Baseline (randomization) and then 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: LS mean change from randomization
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 195 | 191
LS mean change from randomization | -3.70 [-4.31 to -3.09] | -2.46 [-3.08 to -1.84]

13. Secondary Outcome: Least Square Mean Change From Randomization to Week 1 in HAM-A Somatic Anxiety Subscale Score
Description: as for outcome 11
Time Frame: Baseline (randomization) and then 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: LS mean change from randomization
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 195 | 191
LS mean change from randomization | -2.74 [-3.27 to -2.21] | -2.0 [-2.54 to -1.47]

14. Secondary Outcome: Least Square Mean Change From Randomization to Week 1 in CGI-S Score
Description: Results based on MITT population with available data for this outcome measure.
Time Frame: Baseline (randomization) and then 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: LS mean change from randomization
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 195 | 191
LS mean change from randomization | -0.56 [-0.69 to -0.43] | -0.35 [-0.48 to -0.22]

15. Secondary Outcome: Number of Patients With HAM-A Response (≥50% Score Reduction From Randomization) at Week 1
Description: as for outcome 11
Time Frame: Baseline (randomization) and then 8 weeks
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 195 | 191
Participants | 33 | 22

ADVERSE EVENTS:
Arm/Group | Quetiapine XR | Placebo
Serious Adverse Events (participants affected / at risk) | 0/209 | 0/200
Other Adverse Events (participants affected / at risk) | 154/209 | 120/200
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine XR (N=209) | Placebo (N=200)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 3 | 1
Sinus Arrhythmia (Cardiac disorders) | 0 | 1
Supraventricular Extrasystoles (Cardiac disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Blepharitis (Eye disorders) | 0 | 1
Blepharospasm (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 2 | 0
Dry Eye (Eye disorders) | 0 | 1
Vision Blurred (Eye disorders) | 2 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 2
Abnormal Faeces (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 13 | 8
Diarrhoea (Gastrointestinal disorders) | 6 | 6
Dry Mouth (Gastrointestinal disorders) | 49 | 16
Dyspepsia (Gastrointestinal disorders) | 6 | 3
Flatulence (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 12 | 12
Stomach Discomfort (Gastrointestinal disorders) | 2 | 0
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 3
Chest Discomfort (General disorders) | 1 | 2
Chest Pain (General disorders) | 2 | 0
Fatigue (General disorders) | 20 | 8
Gait Disturbance (General disorders) | 1 | 0
Irritability (General disorders) | 4 | 1
Malaise (General disorders) | 1 | 0
Oedema (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Sluggishness (General disorders) | 1 | 0
Thirst (General disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Seasonal Allergy (Immune system disorders) | 3 | 0
Breast Infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Conjunctivitis Infective (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Enterobiasis (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 4 | 2
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 7 | 17
Otitis Externa (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 1
Rhinovirus Infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 5 | 4
Tooth Abscess (Infections and infestations) | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 5
Urinary Tract Infection (Infections and infestations) | 4 | 2
Viral Infection (Infections and infestations) | 1 | 1
Joint Sprain (Injury, poisoning and procedural complications) | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Blood Cholesterol Increased (Injury, poisoning and procedural complications) | 1 | 0
Blood Prolactin Increased (Injury, poisoning and procedural complications) | 0 | 1
Blood Triglycerides Increased (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram QT Prolonged (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram T Wave Amplitude Decreased (Injury, poisoning and procedural complications) | 1 | 0
Glycosylated Haemoglobin Increased (Injury, poisoning and procedural complications) | 1 | 1
Lipids Increased (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil Count Decreased (Injury, poisoning and procedural complications) | 1 | 0
Weight Decreased (Injury, poisoning and procedural complications) | 0 | 2
Weight Increased (Injury, poisoning and procedural complications) | 8 | 2
White Blood Cell Count Decreased (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Increased Appetite (Metabolism and nutrition disorders) | 8 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Contusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 5
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Akathisia (Nervous system disorders) | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0
Balance Disorder (Nervous system disorders) | 1 | 0
Disturbance In Attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 22 | 9
Dysarthria (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 24 | 21
Hypersomnia (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 1
Lethargy (Nervous system disorders) | 3 | 0
Migraine (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 5 | 1
Psychomotor Hyperactivity (Nervous system disorders) | 2 | 1
Restless Legs Syndrome (Nervous system disorders) | 2 | 0
Sedation (Nervous system disorders) | 26 | 5
Somnolence (Nervous system disorders) | 47 | 24
Speech Disorder (Nervous system disorders) | 0 | 1
Tension Headache (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 3 | 1
Abnormal Dreams (Psychiatric disorders) | 6 | 2
Agitation (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Crying (Psychiatric disorders) | 1 | 0
Depressed Mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 3 | 3
Generalised Anxiety Disorder (Psychiatric disorders) | 0 | 2
Initial Insomnia (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 15 | 3
Libido Decreased (Psychiatric disorders) | 5 | 0
Nightmare (Psychiatric disorders) | 2 | 1
Restlessness (Psychiatric disorders) | 3 | 1
Sleep Disorder (Psychiatric disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0
Ejaculation Delayed (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Sebaceous Cyst Excision (Vascular disorders) | 1 | 0
Hot Flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 1
Orthostatic Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If Sponsor does not publish within 2 years after study completion, PI is permitted to publish, with confidential information removed from manuscript. Sponsor will have opportunity to review and approve publication at least 60 days prior to being submitted/disclosed. Sponsor can request, in writing, an additional 90 day embargo.